CLINICAL TRIAL: NCT03505372
Title: Role of Contrast Enhanced Spectral Mammography to Predict Upgrade Rates of Biopsy Proven Atypical Ductal Hyperplasia
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Unable to recruit to study due to limited number of patients with ADH
Sponsor: Dana-Farber Cancer Institute (Other)
Collaborators: GE Healthcare (Industry)
Responsible Party: Principal Investigator, Jordana Phillips, MD, Principal Investigator, Dana-Farber Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 17-694
Record Dates: First submitted 2018-04-04; First posted 2018-04-23 (Actual); Results first posted 2020-02-11 (Actual); Last update posted 2020-02-11 (Actual); Status verified 2020-01

CONDITIONS: Atypical Ductal Hyperplasia
Keywords: Atypical ductal hyperplasia; ADH
MeSH Terms: conditions — Carcinoma, Intraductal, Noninfiltrating

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: No

ARMS (1):
- Contrast enhanced mammography (Experimental): * The CESM images will be performed according to clinical protocol
  * Images will be acquired within approximately 2-12 minutes of contrast injection
  * A total of four images per breast will be acquired with low and high energy
  * Two radiologists will prospectively review the CESM, and will use a third as tie-breaker
  * The CESM will be evaluated for the biopsy site and up to two additional findings in either breast
  * The biopsy site will be evaluated for abnormal findings that would suggest malignant involvement
  Interventions: Device: Contrast enhanced mammography

INTERVENTIONS:
Device: Contrast enhanced mammography — Contrast enhanced mammography is a new type of mammogram that uses contrast material combined with the mammogram to highlight areas that might be breast cancer and that could be missed on the mammogram alone.

SUMMARY:
This research study is studying whether contrast enhanced mammography can predict if atypical ductal hyperplasia will progress to cancer.

The device involved in this study is:

-Contrast enhanced mammography

DETAILED DESCRIPTION:
This research study is a Pilot Study, which is the first time investigators are examining this study device for this purpose.

Atypical ductal hyperplasia (ADH) is a common diagnosis after breast biopsy. Although it is not cancer itself, ADH can become breast cancer in some cases. As a result, surgery is performed to remove ADH to make sure it doesn't progress to cancer. In many cases, no cancer is found during the surgery.

Previous studies have shown that breast MRI may be able to predict which areas of ADH will be cancer at the time of surgery. This would help prevent unnecessary surgery in some patients.

Contrast enhanced mammography is a new type of mammogram that is already being used in clinical practice to help find breast cancer. Similar to breast MRI, it uses contrast material combined with the mammogram to highlight areas that might be breast cancer and that could be missed on the mammogram alone. Contrast material is a dye or other substance that helps show abnormal areas within the body.

Studies have shown the contrast enhanced mammography has a similar ability to find breast cancer as breast MRI.

The investigators purpose is to see whether contrast enhanced mammography can predict which areas of ADH will become breast cancer at the time of surgery. The investigators believe this will help prevent unnecessary surgery in many with women with the diagnosis of ADH.

ELIGIBILITY:
Inclusion Criteria:

* Age, Minimum 30 years. CESM is an imaging exam that uses radiation and is not typically employed in women younger than age 30 due to potentially negative biologic effects on glandular breast tissue.
* Participants who had a percutaneous breast biopsy (to include stereotactic, tomosynthesis, or ultrasound guided) that revealed ADH
* Participants will be undergoing surgical excision to remove the ADH.
* Participants must have normal organ and marrow function as defined by a GFR ≥60 mL/min/1.73 m2 to be performed per clinical protocol
* Patients ≥65 years without underlying renal insufficiency get GFR tested within 6 months of the exam.
* Patients < 65 years without underlying renal insufficiency do not require an GFR calculation)
* Patients ≥65 years with known underlying renal insufficiency get GFR tested within 1 month of the exam.
* Patients < 65 years with known renal insufficiency get GFR tested within 1 month of the exam.
* Because of the potential teratogenic effects of radiation, women of child-bearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry, until the CESM is performed. Should a woman become pregnant or suspect she is pregnant, she should inform the study team prior to getting the CESM.
* Ability to understand and the willingness to sign a written informed consent document

Exclusion Criteria:

* Participants with a core biopsy diagnosis of atypia with associated malignancy (in the same quadrant) will be excluded.
* Participant had a breast MRI that was performed after the diagnosis of ADH but before surgical excision
* Participants who have a known allergy to contrast media.
* Participants who have a known severe allergic response to one or more allergens, as defined by anaphylaxis.
* Participants with persistent asthma as defined by the National Heart, Lung, and Blood Institute.
* Participants with renal insufficiency or failure, as determined by a point of care renal function blood test.
* Participants who are breastfeeding are excluded because there is an unknown but potential risk for adverse events in nursing infants secondary to contrast administration in the mother.
* Participants with the following underlying medical conditions: multiple myeloma, myasthenia gravis, dysproteinemias, severe cardiac disease, aortic stenosis, primary pulmonary hypertension, cardiac arrythmia, or severe cardiomyopathy. These underlying medical conditions may make the participant more likely to develop a contrast reaction. This is based on the ACR contrast manual version 10.3 and hospital policy.
* Participants with thyroid carcinoma or thyroid disease for whom systemic radioactive iodine therapy is part of planned diagnostic work-up or treatment within 2 months following the contrast mammogram study.
* Participants with a concurrent active illness including, but not limited to, symptomatic congestive heart failure, unstable angina pectoris, cardiac arrhythmia, thyroid storm.
* Pregnant women are excluded from this study because CESM uses radiation with the potential for teratogenic or abortifacient effects. This will be defined by a urine pregnancy test prior to the CESM study.

Min Age: 30 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 5 (Actual)
Dates: Start 2018-05-10 (Actual); Primary Completion 2019-06-28 (Actual); Study Completion 2019-06-28 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Jordana Phillips, MD, Principal Investigator — Beth Israel Deaconess Medical Center
Locations (1):
- Beth Israel Deaconess Medical Center, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 5 patients were recruited
Groups:
- Contrast Enhanced Mammography: * The CESM images will be performed according to clinical protocol
  * Images will be acquired within approximately 2-12 minutes of contrast injection
  * A total of four images per breast will be acquired with low and high energy
  * Two radiologists will prospectively review the CESM, and will use a third as tie-breaker
  * The CESM will be evaluated for the biopsy site and up to two additional findings in either breast
  * The biopsy site will be evaluated for abnormal findings that would suggest malignant involvement
  Contrast enhanced mammography: Contrast enhanced mammography is a new type of mammogram that uses contrast material combined with the mammogram to highlight areas that might be breast cancer and that could be missed on the mammogram alone.
Period: Overall Study
Arm/Group | Contrast Enhanced Mammography
Started | 5
Completed | 5
Not Completed | 0

BASELINE CHARACTERISTICS:
Population: Patients who had ADH and were getting surgical excision were enrolled. We terminated the study as recruitment was too low to continue.
Arm/Group | Contrast Enhanced Mammography
Number analyzed (Participants) | 5
Age, Categorical [Count of Participants; unit: Participants] — > or = to 30 years old
  Participants
    <=18 years | 0
    Between 18 and 65 years | 5
    >=65 years | 0
Age, Continuous [Mean (Full Range); unit: years] | 50.2 [47 to 56]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5
  Male | 0
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 5

OUTCOME MEASURES:

1. Primary Outcome: CESM's Ability to Predict Upgrade Rates of Biopsy Proven ADH at Surgical Excision
Description: Investigators will evaluate whether enhancement on CESM can predict which cases of ADH upgrade at the time of surgical excision.
Time Frame: 3 months
Population: Images were performed but outcome data was not collected and therefore we cannot provide any analysis.
Arm/Group | Contrast Enhanced Mammography
Number analyzed (Participants) | 0

2. Secondary Outcome: Types of Changes in Surgical Management Based on CESM
Description: Investigators will evaluate how incidental findings seen on CESM impact the surgical management of patients diagnosed with ADH. The initial surgical management documented in the clinical report (created before CESM performed) will be compared with the surgical management documented in the medical record after the CESM was performed to determine the change.
Time Frame: 3 months
Population: Images were performed but outcome data was not collected and therefore we cannot provide any analysis.
Arm/Group | Contrast Enhanced Mammography
Number analyzed (Participants) | 0

ADVERSE EVENTS:
Time Frame: 3 months
Arm/Group | Contrast Enhanced Mammography
All-Cause Mortality (participants affected / at risk) | 0/5
Serious Adverse Events (participants affected / at risk) | 0/5
Other Adverse Events (participants affected / at risk) | 0/5

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-12-09): https://cdn.clinicaltrials.gov/large-docs/72/NCT03505372/Prot_SAP_000.pdf